CLINICAL TRIAL: NCT01869972
Title: Biological Variation of Phenylalanine in Patients With Hyperphenylalaninemia
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster Children's Hospital (Other); Children's Hospital of Eastern Ontario (Other); BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: PKUvar-01
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Phenylketonuria; Hyperphenylalaninemia
Keywords: PKU; phenylketonuria; hyperphenylalaninemia; Kuvan; sapropterin
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Wide PHE group: Subjects prescribed diet alone to treat their PKU who have >1/3 of monitoring phenylalanine levels (with at least 3 levels measured) outside the target treatment range in the 6 months preceding enrolment. Target therapeutic range is 120 - 360 umol/L for age <12 years and 120 - 600 umol/L for age ≥ 12 years.
- Target PHE group: Subjects prescribed diet alone to treat their PKU who have ≤ 1/3 of monitoring phenylalanine levels (with at least 3 levels measured) outside the target treatment range in the 6 months preceding enrolment. Target therapeutic range is 120 - 360 umol/L for age <12 years and 120 - 600 umol/L for age ≥ 12 years.
- Kuvan(TM) group: Subjects on Kuvan(TM) (any dose for at least 3 months with no dosage change for most recent 1 month) ± diet therapy
- Control group: Subjects with non-PKU hyperphenylalaninemia (maximum phenylalanine level 120 - 599 umol/L on no therapy).

SUMMARY:
Phenylketonuria (PKU) is a rare disease where the level of phenylalanine (one of the amino acids) in the body is greatly increased. High levels can cause brain damage, especially in babies and children. This brain damage can be prevented if a special low phenylalanine diet is started soon after birth. A new drug, sapropterin, can also lower phenylalanine levels in some patients. PKU therapy is monitored by measuring the blood phenylalanine every week, with the goal to keep the level within a target range. Recently, studies have suggested that the variation in the blood phenylalanine may be just as important as the absolute blood phenylalanine level for brain outcome.

The investigators will look at the variation in blood phenylalanine level over 24 hours to see how much the level changes. The investigators will measure this in patients with typical PKU who are compliant with the diet and in patients who are not compliant with the diet. The investigators will also measure this in patients with "mild" PKU who do not usually have as high levels of phenylalanine. Finally, the investigators will see if patients on sapropterin have lower variation.

DETAILED DESCRIPTION:
Phenylketonuria (OMIM 261600) results from the inherited deficiency of the enzyme phenylalanine hydroxylase, (PAH, Enzyme Classification 1.14.16.1). A deficiency of this enzyme leads to elevated blood and tissue levels of the amino acid phenylalanine upon exposure to normal amounts of dietary protein. The elevated phenylalanine in the brain is harmful to cognitive development, usually resulting in permanent severe mental retardation. Soon after the development of a special dietary treatment for PKU and of a simple screening test to detect elevated phenylalanine, newborn screening for PKU became widespread and early detection and treatment largely prevented the severe neurological effects of PKU.

With population-based detection of hyperphenylalaninemia, it soon became apparent that there was significant biological variation of phenylalanine levels between patients (i.e. inter-individual biological variation) with phenylketonuria (PKU) and this now forms part of the classification system for hyperphenylalaninemia (i.e. benign hyperphenylalaninemia, mild, moderate or classical phenylketonuria). While variations of the classification system exist, most commonly "classical" PKU refers to individuals with plasma phenylalanine levels greater than 1200 µmol/L on an unrestricted diet. "Moderate" PKU refers to levels between 900 and 1200 µmol/L, while "mild" PKU refers to levels between 600 and 900 µmol/L. "Non-PKU" or "benign" hyperphenylalaninemia refers to phenylalanine levels less than 600 µmol/L on an unrestricted diet, that while greater than normal phenylalanine levels (< 100 µmol/L), historically have not been prescribed dietary restriction of phenylalanine. This inter-individual variation is generally due to variable residual enzyme activity and genotype in PKU patients.

Intra-individual variation (the changes of phenylalanine levels in one individual) has been observed by all clinicians who treat PKU. While some of this variation is simply the expression of the underlying genotype when a patient's dietary phenylalanine level exceeds prescribed amounts (i.e. "cheating" on their diet), other variation represents shifts from anabolic to catabolic states in a diurnal pattern or during intercurrent illness. While overall exposure to high phenylalanine has long been known to adversely affect IQ scores, recently increased variability in phenylalanine levels has been reported to be linked to lower IQ, highlighting the importance of improving our understanding of intra-individual variation.

New treatments for PKU, therefore, need to be assessed in terms of their effect on biological variation of phenylalanine. Sapropterin dihydrochloride (KuvanTM) is a small molecule drug that can lower phenylalanine levels in patients with phenylalanine hydroxylase deficiency by a direct interaction with the enzyme . The pharmacokinetics of KuvanTM have been evaluated in adults and are undergoing evaluation in pediatric patients, however, the biological effect of KuvanTM in terms of lowering of blood phenylalanine levels would be expected to have a longer profile than the blood levels of the drug itself because the half-life of the activated enzyme would be longer. This suggests that KuvanTM may have a modulating effect on variation of blood phenylalanine levels in PKU patients.

In this observational study, the investigators will directly measure the short-term biological variation of blood phenylalanine in hyperphenylalaninemic patients by frequent measurements of phenylalanine levels over a 24 hour period. The investigators will enroll subjects already followed at one of the two study sites who are treated by diet alone or who are treated with KuvanTM therapy (+/- diet). During the 24 hour period subjects will be asked to maintain their typical diet/therapy.

Hypothesis: Biological variation will be less in KuvanTM treated patients than in classical phenylketonuria treated by diet alone.

OBJECTIVES:

Determine short-term biologic variation in people with hyperphenylalaninemia, with and without KuvanTM therapy.

ELIGIBILITY:
Inclusion Criteria:

• Subjects ≥4 years of age with hyperphenylalaninemia. Must have at least 1 documented blood phenylalanine level >600 µmol/L for study groups (Wide PHE, Target PHE, Kuvan groups) or >120 µmol/L for control group.

Exclusion Criteria:

* Significant cognitive impairment (IQ <70 or clinical judgment).
* Pregnancy
* Other specific PKU therapies, including enzyme replacement therapy or any amino acid supplement designed to block uptake or transport of phenylalanine (i.e. large neutral amino acid mixtures)
* Any intercurrent illness within the previous 5 days (any of fever, vomiting, diarrhea, decreased intake, upper respiratory tract infection).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metabolic and/or PKU clinic
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Standard deviation of blood phenylalanine level (sdPHE) | 24 hour period
  16 to 17 blood phenylalanine levels will be measured over 24 hours. The standard deviation of those measurements will be the sdPHE.

SECONDARY OUTCOMES:
Peak phenylalanine level | 24 hour
  The highest blood phenylalanine level in the 24 hour period
peak phenylalanine / tyrosine ratio | 24 hours
  The highest blood phenylalanine / tyrosine ratio, with phenylalanine and tyrosine measured on the same sample

CONTACTS AND LOCATIONS:
Overall Officials: Murray Potter, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario